CLINICAL TRIAL: NCT05637424
Title: Potential of Urine Biomarkers CHI3L1, NGAL, TIMP-2, IGFBP7 and Combinations as Complementary Diagnostic Tools for Acute Kidney Injury After Pediatric Cardiac Surgery: a Prospective Cohort Study
Brief Title: Urine Biomarkers to Predict Acute Kidney Injury After Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201213147
Record Dates: First submitted 2022-11-17; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury; Congenital Cardiac Disorders
Keywords: acute kidney injury; pediatric; cardiac surgery; biomarkers
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood samples were taken. Volume and number of blood samples collected were according to the guidance of the European Commission on blood volume limits for sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort study is to evaluate, in pediatric patients after cardiac surgery, the predicting capability of biomarkers for acute kidney injury. The main questions it aims to answer:

* The predicting capability of acute kidney injury (AKI) biomarkers for the primary endpoint: the occurrence of AKI stage ≥ 1 within 48-h after intensive care unit (ICU) admission.
* The predicting capability of AKI biomarkers for the secondary endpoint: the occurrence of AKI stage ≥ 2 within 12-h after ICU admission.
* Investigated biomarkers include urine chitinase 3-like protein 1 (uCHI3L1), urine neutrophil gelatinase-associated lipocalin (uNGAL), tissue inhibitor of metalloproteinases-2 (TIMP-2), insulin-like growth factor-binding protein 7(IGFBP7), NephroCheck® and Δ serum creatinine [postop-preop]. Differences in concentration between patients with and without AKI development were investigated, as well as AKI diagnostic performance of (combined) biomarkers.

During and after cardiac surgery several blood and urine samples will be taken of participants to investigated AKI occurrence and to measure biomarker concentrations.

DETAILED DESCRIPTION:
Pediatric patients after cardiac surgery were prospectively included. Urine and blood samples were taken between induction of anesthesia and the start of cardiac surgery, at intensive care unit (ICU) admission and 2, 4, 6, 12, 24, 48-h after ICU admission respectively.

Sampling was only done in the operating room and ICU. Volume and number of blood samples collected were according to the guidance of the European Commission on blood volume limits for sampling. Clinical data were extracted from the hospital records by study coordinators. Samples were anonymized as were clinical data. All technicians were blinded to clinical data.

Acute kidney injury was defined by the Kidney Disease Improving Global Outcomes (KDIGO) definition and classification, using both serum creatine as urine output criteria. AKI predicting capability of biomarkers was assessed by performing area under the receiver-operating characteristics curve (AUROC) analysis. Biomarkers were evaluated individual and as a combination of two- or three-biomarker-panels diagnostic tests. Additionally, the absolute difference between pre- and postoperative serum creatinine (ΔsCr[postop-preop]) was evaluated as diagnostic test.

To correct for urine dilution, the investigated urine biomarkers were normalized, by dividing urine biomarker concentration by urine creatinine concentration.

A sensitivity analysis was made to evaluate the biomarker performance to predict AKI ≥ 1 in patients who did not already have AKI ≥ 1 at ICU admission. Likewise, a similar sensitivity analysis was made for AKI ≥ 2.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (age <18 years with body weight ≥ 2 kg)
* patient underwent elective cardiac surgery

Exclusion Criteria:

* AKI stage ≥1 on admission
* chronic kidney disease (CKD) stage 5
* kidney transplantation
* cardiac surgery during weekend

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients (age <18 years with body weight ≥ 2 kg) who underwent elective cardiac suregry, prospective enrolled preoperatively at Ghent University hospital. Exclusion criteria were AKI stage ≥1 on admission, chronic kidney disease (CKD) stage 5, kidney transplantation, surgery during weekend
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
AKI stage ≥ 1 | 48 hours after ICU admission
  occurrence of AKI stage ≥ 1 within 48 hours after ICU admission after pediatric cardiac surgery

SECONDARY OUTCOMES:
AKI stage ≥ 2 | 12 hours after ICU admission
  occurrence of AKI stage ≥ 2 within 12 hours after ICU admission after pediatric cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, M.D.; Ph.D., Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918